CLINICAL TRIAL: NCT04166058
Title: A Phase 3, Open-label, Long-term Safety Study of Oral Linaclotide Administered to Pediatric Participants With Functional Constipation (FC) or Irritable Bowel Syndrome With Constipation (IBS-C)
Brief Title: Long-term Safety of Linaclotide in Pediatric Participants With FC or IBS-C
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AbbVie (Industry)
Collaborators: Ironwood Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LIN-MD-66; 2019-001955-38 (EudraCT Number)
Record Dates: First submitted 2019-11-11; First posted 2019-11-18 (Actual); Results first posted 2026-01-06 (Actual); Last update posted 2026-01-06 (Actual); Status verified 2025-11

CONDITIONS: Irritable Bowel Syndrome With Constipation; Functional Constipation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- 72 μg linaclotide (Active Comparator): An oral capsule that is taken once daily. It may be taken whole or sprinkled into 1 teaspoonful of applesauce or 30mL of bottled water.
  Interventions: Drug: Functional Constipation (FC) participants (LIN-MD-62 and LIN-MD-64 completers)
- 145 μg linaclotide (Active Comparator): An oral capsule that is taken once daily. It may be taken whole or sprinkled into 1 teaspoonful of applesauce or 30mL of bottled water.
  Interventions: Drug: Irritable Bowel Syndrome with Constipation (IBS-C) participants (LIN-MD-63 and LIN-MD-64 completers); Drug: Functional Constipation (FC) participants (LIN-MD-62 and LIN-MD-64 completers)
- 290 μg linaclotide (Active Comparator): An oral capsule that is taken once daily. It may be taken whole or sprinkled into 1 teaspoonful of applesauce or 30mL of bottled water.
  Interventions: Drug: Irritable Bowel Syndrome with Constipation (IBS-C) participants (LIN-MD-63 and LIN-MD-64 completers)

INTERVENTIONS:
Drug: Irritable Bowel Syndrome with Constipation (IBS-C) participants (LIN-MD-63 and LIN-MD-64 completers) — Participants who completed study LIN-MD-63 at their time of enrollment will be assigned a dose of 290 μg. Participants who received ≤ 145 μg linaclotide or placebo in study LIN-MD-63 at the time of completion will continue to receive 145 μg.
  Participants who completed study LIN-MD-64 at their time of enrollment will be assigned a dose of 290 μg if they choose to receive open-label or continue to receive blinded dose of 145 or 290 μg if they choose to remain on the same blinded dose.
  Arms: 145 μg linaclotide; 290 μg linaclotide
Drug: Functional Constipation (FC) participants (LIN-MD-62 and LIN-MD-64 completers) — Participants whom are between the ages of 6-11 years old at their time of enrollment will be assigned a dose of 72 μg.
  Participants whom are between the ages of 12-17 years old at their time of enrollment will be randomized at 1:1 ratio to 72 or 145 μg linaclotide.
  Arms: 145 μg linaclotide; 72 μg linaclotide

SUMMARY:
LIN-MD-66 is a Phase 3 open-label study with 24 weeks (Functional Constipation participants) or 52 weeks (Irritable bowel syndrome with constipation participants) of linaclotide exposure that will enroll pediatric participants (6-17 years of age) with FC or IBS-C who completed study intervention in studies LIN-MD-62, LIN-MD-63, or LIN-MD-64 based on the individual study criteria.

ELIGIBILITY:
Inclusion Criteria:

* Participant weighs ≥ 18 kg at the time the parent/guardian/LAR and/or caregiver has provided signed consent.
* Female participants who have had their first menstrual period and are sexually active must agree to use a reliable form of contraception.
* Participants must have completed study intervention in their lead-in study.

Inclusion Criteria for Phase 2 LIN-MD-62 or Phase 2 LIN-MD-63 and Phase 3 LIN-MD-64 completers who enroll in LIN-MD-66 after >28 days from last study intervention:

- Female participants of childbearing potential must have a negative serum pregnancy test at the Screening Visit (Visit 1) and negative urine pregnancy test prior to the first dose on the Day 1 Visit (Visit 2).

Exclusion Criteria:

* Participant has a known allergy or sensitivity to the study intervention or its components or other medications in the same drug class.
* Participant received an investigational drug, other than linaclotide, during the 30 days before the Screening Visit (Visit 1) or is planning to receive an investigational drug (other than that administered during this study) or use an investigational device at any time during the study.
* Female participants who are currently pregnant or nursing, or plan to become pregnant or nurse during the clinical study.
* Participant has required manual disimpaction any time prior to study intervention or disimpaction during in-patient hospitalization within 1 year prior to study intervention.
* Participant has any of the following conditions:

  * a) Down's syndrome or any other chromosomal disorder
  * b) Anatomic malformations (eg, imperforate anus, anal stenosis, anterior displaced anus)
  * c) Intestinal nerve or muscle disorders (eg, Hirschprung disease, visceral myopathies, visceral neuropathies)
  * d) Neuropathic conditions (eg, spinal cord abnormalities, neurofibromatosis, tethered cord, spinal cord trauma)
  * e) Neurodevelopmental disabilities (early-onset, chronic disorders that share the essential feature of a predominant disturbance in the acquisition of cognitive, motor, language, or social skills, which has a significant and continuing impact on the developmental progress of an individual) producing a cognitive delay that precludes comprehension by the participant.
* Participant has a mechanical bowel obstruction or pseudo-obstruction.
* Participant currently has both unexplained and clinically significant alarm symptoms (lower GI bleeding [rectal bleeding or heme-positive stool], iron-deficiency anemia, or any unexplained anemia, or weight loss) and systemic signs of infection or colitis, or any neoplastic process.
* Participant has an active anal fissure (Note: history of anal fissure is not an exclusion).
* Participant has had surgery that meets any of the following criteria:

  * a) Bariatric surgery for treatment of obesity, or surgery to remove a segment of the GI tract at any time before the Screening Visit (Visit 1).
  * b) Surgery of the abdomen, pelvis, or retroperitoneal structures during the 6 months before the Screening Visit (Visit 1)
  * c) An appendectomy or cholecystectomy during the 60 days before the Screening Visit
  * d) Other major surgery during the 30 days before the Screening Visit (Visit 1)
* Participant is receiving enteral tube feeding
* Participants who have positive urine drug screen results for cocaine, barbiturates, opiates, or cannabinoids will be excluded from study participation.

Exclusion Criteria for LIN-MD-62, LIN-MD-63 and LIN-MD-64 Completers Who Enroll in LIN-MD-66 > 28 Days From Last Study Intervention:

* Participant has a history of nonretentive fecal incontinence
* Participant has a history of drug or alcohol abuse
* Participant has any of the following conditions:

  * a) Celiac disease, or positive serological test for celiac disease and the condition has not been ruled out by endoscopic biopsy
  * b) Cystic fibrosis
  * c) Hypothyroidism that is untreated or treated with thyroid hormone at a dose that has not been stable for at least 3 months prior to the Screening (Visit 1)
  * d) Lead toxicity, hypercalcemia
  * e) Inflammatory bowel disease
  * f) Childhood functional abdominal pain syndrome
  * g) Childhood functional abdominal pain
  * h) Poorly treated or poorly controlled psychiatric disorders that might influence his or her ability to participate in the study
  * i) Lactose intolerance that is associated with abdominal pain or discomfort and could confound the assessments in this study
  * j) History of cancer other than treated basal cell carcinoma of the skin. (Note: Participants with a history of cancer are allowed provided that the malignancy has been in a complete remission for at least 5 years before the Randomization Visit. A complete remission is defined as the disappearance of all signs of cancer in response to treatment.)
  * k) History of diabetic neuropathy
* Participants who have positive urine drug screen results for cocaine, barbiturates, opiates, or cannabinoids.

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 381 (Actual)
Dates: Start 2019-11-19 (Actual); Primary Completion 2025-06-05 (Actual); Study Completion 2025-06-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: ABBVIE INC., Study Director — AbbVie
Locations (72):
- United States (65):
  - Central Research Associates /ID# 237953, Birmingham, Alabama
  - G & L Research, LLC /ID# 238093, Foley, Alabama
  - The Center for Clinical Trials Inc. /ID# 234605, Saraland, Alabama
  - HealthStar Research of Hot Springs PLLC /ID# 234608, Hot Springs, Arkansas
  - Preferred Research Partners /ID# 237109, Little Rock, Arkansas
  - Applied Research Center of Arkansas /ID# 238069, Little Rock, Arkansas
  - Advanced Research Center /ID# 237960, Anaheim, California
  - Kindred Medical Institute, LLC /ID# 237367, Corona, California
  - Duplicate_Center for Clinical Trials LLC /ID# 234629, Paramount, California
  - Medical Ctr for Clin Research /ID# 236911, San Diego, California
  - Lynn Institute of Denver /ID# 238086, Aurora, Colorado
  - Childrens National Medical Center /ID# 234417, Washington D.C., District of Columbia
  - Prohealth Research Center /ID# 234659, Doral, Florida
  - Dolphin Medical Research /ID# 234676, Doral, Florida
  - Amedica Research Institute Inc /ID# 234666, Hialeah, Florida
  - Nemours Childrens Specialty Care /ID# 237991, Jacksonville, Florida
  - Elite Clinical Research /ID# 234651, Miami, Florida
  - My Preferred Research LLC /ID# 237943, Miami, Florida
  - South Miami Medical & Research Group Inc. /ID# 234654, Miami, Florida
  - Valencia Medical & Research Center /ID# 234671, Miami, Florida
  - Advanced Research for Health Improvement /ID# 238253, Naples, Florida
  - Pediatric & Adult Research Center /ID# 234681, Orlando, Florida
  - Nemours Children's Hospital /ID# 234429, Orlando, Florida
  - Oviedo Medical Research /ID# 234692, Oviedo, Florida
  - Treken Primary Care /ID# 234645, Atlanta, Georgia
  - Children's Healthcare of Atlanta - Ferry Rd /ID# 237005, Atlanta, Georgia
  - Children's Ctr Digestive, US /ID# 237574, Atlanta, Georgia
  - River Birch Research Alliance /ID# 237963, Blue Ridge, Georgia
  - Clinical Research Institute /ID# 234702, Stockbridge, Georgia
  - Sleep Care Research Institute d/b/a Clinical Research Institute /ID# 236342, Stockbridge, Georgia
  - KU Wichita Center for Clinical Research /ID# 234500, Wichita, Kansas
  - Michael W. Simon, MD, PSC /ID# 236516, Lexington, Kentucky
  - Virgo Carter Pediatrics /ID# 234518, Silver Spring, Maryland
  - MNGI Digestive Health, P. A. /ID# 234437, Minneapolis, Minnesota
  - GI associates and Endoscopy Ce /ID# 237969, Flowood, Mississippi
  - David M. Headley, MD, P.A. /ID# 238216, Port Gibson, Mississippi
  - Private Practice - Dr. Craig Spiegel /ID# 234545, Bridgeton, Missouri
  - Medclinical Research Partners LLC/ Foundation Pediatrics /ID# 234566, East Orange, New Jersey
  - University of New Mexico /ID# 236983, Albuquerque, New Mexico
  - Columbia University Irving Medical Center /ID# 235686, New York, New York
  - Advantage Clinical Trials /ID# 237932, The Bronx, New York
  - East Carolina University - Brody School of Medicine /ID# 237509, Greenville, North Carolina
  - PMG Research of Piedmont Healthcare-Statesville /ID# 238257, Statesville, North Carolina
  - Univ Oklahoma HSC /ID# 237546, Oklahoma City, Oklahoma
  - IPS Research Company /ID# 237669, Oklahoma City, Oklahoma
  - Frontier Clinical Research, LLC - Scottdale /ID# 238022, Scottdale, Pennsylvania
  - Duplicate_Frontier Clinical Research /ID# 237923, Smithfield, Pennsylvania
  - Rhode Island Hospital /ID# 237861, Providence, Rhode Island
  - Coastal Pediatric Research - West Ashley B /ID# 234678, Charleston, South Carolina
  - Coastal Pediatric Research - Summerville /ID# 234674, Summerville, South Carolina
  - The Jackson Clinic, PA /ID# 236772, Jackson, Tennessee
  - Accellacare of Knoxville /ID# 234462, Jefferson City, Tennessee
  - Cook Children's Med. Center /ID# 237536, Fort Worth, Texas
  - Valley Institute of Research /ID# 234475, Harlingen, Texas
  - Vilo Research Group Inc /ID# 238228, Houston, Texas
  - Cullen Research /ID# 234482, Houston, Texas
  - Pioneer Research Solutions - Houston /ID# 236935, Houston, Texas
  - AIM Trials /ID# 236364, Plano, Texas
  - Sun Research Institute /ID# 236932, San Antonio, Texas
  - ClinPoint Trials /ID# 236615, Waxahachie, Texas
  - Duplicate_Chrysalis Clinical Research /ID# 234515, St. George, Utah
  - Office of Maria Ona /ID# 234539, Franklin, Virginia
  - Health Research of Hampton Roads, Inc. (HRHR) /ID# 237252, Newport News, Virginia
  - Clinical Research Partners, LLC /ID# 237158, Richmond, Virginia
  - Duplicate_Multicare Institute for Research and Innovation /ID# 236979, Tacoma, Washington
- Canada (3):
  - London Health Sciences Center- University Hospital /ID# 234309, London, Ontario
  - Bluewater Clinical Research Group Inc /ID# 234618, Sarnia, Ontario
  - Stouffville Medical Centre /ID# 234619, Stouffville, Ontario
- Israel (3):
  - Hadassah Hebrew University Hospital - Ein Kerem /ID# 234735, Jerusalem, Jerusalem
  - The Baruch Padeh Medical Center Poriya /ID# 234768, Tiberias, Northern District
  - The Chaim Sheba Medical Center /ID# 236760, Ramat Gan, Tel Aviv
- Duplicate_Academisch Medisch Centrum /ID# 237116, Amsterdam, North Holland, Netherlands

IPD SHARING:
Plan to Share IPD: Yes
AbbVie is committed to responsible clinical trial data sharing. This includes access to anonymized, individual and trial-level data (analysis data sets), as well as other information.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: For details on when studies are available for sharing visit https://vivli.org/ourmember/abbvie/
Access Criteria: To learn more about the process, or to submit a request, visit the following link https://www.abbvieclinicaltrials.com/hcp/data-sharing/
URL: https://vivli.org/ourmember/abbvie/

RESULTS

PARTICIPANT FLOW:
Groups:
- FC 72 ug Linaclotide: Functional Constipation (FC) participants who completed lead-in studies LIN-MD-62 or LIN-MD-64 were dosed as follows in this study:
  Participants aged 6 to 11 years received an open-label dose of linaclotide 72 ug, oral capsule, once daily for 24 weeks.
  Participants aged 12 to 17 years were randomized to receive an open-label dose of linaclotide either 72 or 145 ug, oral capsule, once daily for 24 weeks.
- FC 145 ug Linaclotide: Functional Constipation (FC) participants who completed lead-in studies LIN-MD-62 or LIN-MD-64 were dosed as follows in this study:
  Participants aged 12 to 17 years were randomized to receive an open-label dose of linaclotide either 72 or 145 ug, oral capsule, once daily for 24 weeks.
- IBS-C 145 ug Linaclotide: Irritable Bowel Syndrome with Constipation (IBS-C) participants were dosed as follows:
  Participants who received ≤ 145 ug linaclotide or placebo in lead-in study LIN-MD-63, in this study received an open-label dose of linaclotide 145 ug, oral capsule, once daily for 52 weeks.
  Participants who completed lead-in study LIN-MD-64, in this study had the option to either remain on the same blinded linaclotide dose they were receiving in lead-in study LIN-MD-64 (145 or 290 ug) or received an open-label dose of linaclotide 290 ug, oral capsule, once daily for 52 weeks.
- IBS-C 290 ug Linaclotide: Irritable Bowel Syndrome with Constipation (IBS-C) participants were dosed as follows:
  Participants who completed lead-in study LIN-MD-63, in this study received an open-label dose of linaclotide 290 ug, oral capsule, once daily for 52 weeks.
  Participants who completed lead-in study LIN-MD-64, in this study had the option to either remain on the same blinded linaclotide dose they were receiving in lead-in study LIN-MD-64 (145 or 290 ug) or received an open-label dose of linaclotide 290 ug, oral capsule, once daily for 52 weeks.
Period: Overall Study
Arm/Group | FC 72 ug Linaclotide | FC 145 ug Linaclotide | IBS-C 145 ug Linaclotide | IBS-C 290 ug Linaclotide
Started | 210 | 73 | 22 | 76
Number of Participants Treated and Received Placebo in lead-in Study | 106 | 31 | 2 | 4
Completed | 189 | 66 | 20 | 60
Not Completed | 21 | 7 | 2 | 16
Not completed — Adverse Event | 1 | 1 | 0 | 0
Not completed — Withdrawal by Subject | 4 | 4 | 1 | 10
Not completed — Lost to Follow-up | 9 | 2 | 1 | 1
Not completed — Pregnancy | 1 | 0 | 0 | 0
Not completed — Physician Decision | 2 | 0 | 0 | 2
Not completed — Protocol Violation | 1 | 0 | 0 | 0
Not completed — Lack of Efficacy | 2 | 0 | 0 | 0
Not completed — Other | 1 | 0 | 0 | 1
Not completed — Non-compliance with study drug | 0 | 0 | 0 | 2

BASELINE CHARACTERISTICS:
Population: Safety Population: all participants who received at least 1 dose of study intervention (linaclotide) in this extension study. Number analyzed are participants with data available for analyses of the specific category.
Groups:
- Total: Total of all reporting groups
Arm/Group | FC 72 ug Linaclotide | FC 145 ug Linaclotide | IBS-C 145 ug Linaclotide | IBS-C 290 ug Linaclotide | Total
Number analyzed (Participants) | 210 | 73 | 22 | 76 | 381
Age, Continuous [Mean (Standard Deviation); unit: years] | 10.6 (2.96) | 14.2 (1.78) | 13.7 (2.68) | 12.9 (2.98) | 11.89 (3.15)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 115 | 40 | 15 | 45 | 215
  Male | 95 | 33 | 7 | 31 | 166
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 92 | 37 | 8 | 29 | 166
  Not Hispanic or Latino | 118 | 36 | 14 | 47 | 215
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 0 | 0 | 0 | 2
  Asian | 2 | 3 | 0 | 3 | 8
  Native Hawaiian or Other Pacific Islander | 2 | 0 | 0 | 0 | 2
  Black or African American | 59 | 17 | 3 | 19 | 98
  White | 142 | 52 | 18 | 52 | 264
  More than one race | 3 | 1 | 1 | 1 | 6
  Unknown or Not Reported | 0 | 0 | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment-Emergent Adverse Events (TEAEs).
Description: An adverse event (AE) is defined as any untoward medical occurrence in a patient or clinical investigation participant administered a pharmaceutical product which does not necessarily have a causal relationship with this treatment. The investigator assesses the relationship of each event to the use of study drug. A serious adverse event (SAE) is an event that results in death, is life-threatening, requires or prolongs hospitalization, results in a congenital anomaly, persistent or significant disability/incapacity or is an important medical event that, based on medical judgment, may jeopardize the participant and may require medical or surgical intervention to prevent any of the outcomes listed above. Treatment-emergent adverse events/treatment-emergent serious adverse events (TEAEs/TESAEs) are defined as any event that began or worsened in severity on or after the first dose of study drug.
Time Frame: From first dose of study drug until 30 days following last dose of study drug [up to 24 weeks (FC participants) or 52 weeks (IBS-C participants)].
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | FC 72 ug Linaclotide | FC 145 ug Linaclotide | IBS-C 145 ug Linaclotide | IBS-C 290 ug Linaclotide
Number analyzed (Participants) | 210 | 73 | 22 | 76
Participants
  TEAE | 37 | 15 | 4 | 31
  TESAE | 2 | 0 | 0 | 2

ADVERSE EVENTS:
Time Frame: All-cause mortality and adverse event tables include events reported from the time of informed consent to the end of the study. The median time in follow-up (or mean time participants were followed) was 176.0, 177.0, 373.5, and 369.0 days for FC 72 ug linaclotide, FC 145 ug linaclotide, IBS-C 145 ug linaclotide, and IBS-C 290 ug linaclotide, respectively.
Description: All AEs were coded using MedDRA version 27.1 and 28.0 for FC and IBS-C participants, respectively.
Arm/Group | FC 72 ug Linaclotide | FC 145 ug Linaclotide | IBS-C 145 ug Linaclotide | IBS-C 290 ug Linaclotide
All-Cause Mortality (participants affected / at risk) | 0/210 | 0/73 | 0/22 | 0/76
Serious Adverse Events (participants affected / at risk) | 2/210 | 0/73 | 0/22 | 2/76
Other Adverse Events (participants affected / at risk) | 14/210 | 5/73 | 0/22 | 11/76
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | FC 72 ug Linaclotide (N=210) | FC 145 ug Linaclotide (N=73) | IBS-C 145 ug Linaclotide (N=22) | IBS-C 290 ug Linaclotide (N=76)
CONSTIPATION (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
PYELONEPHRITIS (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
POST PROCEDURAL HAEMORRHAGE (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
MIGRAINE (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
DISRUPTIVE MOOD DYSREGULATION DISORDER (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
MENTAL STATUS CHANGES (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
ADENOIDAL HYPERTROPHY (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
NASAL TURBINATE HYPERTROPHY (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
TONSILLAR HYPERTROPHY (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | FC 72 ug Linaclotide (N=210) | FC 145 ug Linaclotide (N=73) | IBS-C 145 ug Linaclotide (N=22) | IBS-C 290 ug Linaclotide (N=76)
DIARRHOEA (Gastrointestinal disorders) | 12 (14) | 5 (5) | 0 (0) | 7 (9)
INFLUENZA (Infections and infestations) | 2 (2) | 0 (0) | 0 (0) | 4 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
AbbVie requests that any investigator or institution that plans on presenting/publishing results disclosure, provide written notification of their request 60 days prior to their presentation/publication. AbbVie requests that no presentation/publication will be instituted until 12 months after a study is completed, or after the first presentation/publication whichever occurs first. A delay may be proposed of a presentation/publication if AbbVie needs to secure patent or proprietary protection.

DOCUMENTS (2):
  • Study Protocol (2021-04-30): https://cdn.clinicaltrials.gov/large-docs/58/NCT04166058/Prot_000.pdf
  • Statistical Analysis Plan (2022-07-19): https://cdn.clinicaltrials.gov/large-docs/58/NCT04166058/SAP_001.pdf